CLINICAL TRIAL: NCT04056221
Title: Effects of Acupuncture on Xerostomia and Xerophthalmia in Sjögren's Syndrome: a Randomized, Double-blinded Clinical Trial
Brief Title: Effects of Acupuncture on Sjögren's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ana Carolina Fragoso Motta, DDS, PhD (Other)
Responsible Party: Sponsor-Investigator, Ana Carolina Fragoso Motta, DDS, PhD, Professor of Oral Diagnosis, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE: 5419
Record Dates: First submitted 2019-03-17; First posted 2019-08-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Sjogren's Syndrome
Keywords: Sjogren's syndrome; xerostomia; xerophthalmia; acupuncture
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia; Xerophthalmia | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Sjogren syndrome's patients will be randomly assigned to either acupuncture (experimental group) at the selected acupoints (R6, E6,E2, Ig4, VC24, TA23, B2) or sham acupuncture (control group), where the needles do not penetrate the skin into non acupuncture points, for 8 weeks, 20 minutes sessions with 12 weeks of follow up.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both patients and investigators who will assess the outcomes have no knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture (Experimental): Acupuncture at the selected points.
  Interventions: Other: Acupuncture
- Sham acupuncture (Sham Comparator): Similar appearance to conventional acupuncture, however, without needles skin penetration.
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture stimulation was done manually, using single-use acupuncture needles that will be inserted on the selected acupoints (R6, E6, E2, Ig4, VC24, TA23, B2) once a week,for 8 weeks, 20 minutes sessions with 12 weeks of follow up.
  Arms: acupuncture
Other: Sham acupuncture — The sham acupuncture consists of needles that achieves no skin penetration and are holden on the points by an adhesive pad.
  Arms: Sham acupuncture

SUMMARY:
Sjögren's syndrome (SS) is a multisystemic chronic autoimmune disease characterized by lymphocytic infiltration of the exocrine glands, resulting in salivary and lacrimal glands hypofunction, with symptoms of dry eyes and mouth. Xerostomia and xerophthalmia present profound negative impact on patients' quality of life, especially due to difficulties in swallowing, dysarthria, dysgeusia, halitosis and burning tongue, discomfort and visual disturbances that lead to daily activities difficulty such as driving or reading. Although some drugs may improve symptoms and prevent SS complications, they can cause significant adverse effects and even fail to relieve symptoms. Integrative and complementary techniques have become a therapeutic option for SS patients. Scientific evidence has supported the efficacy of acupuncture in relieving symptoms of xerostomia and xerophthalmia. Due to the lack of well-controlled and standardized clinical studies, this study aimed to conduct a randomized and controlled trial to determine the efficacy of acupuncture as a therapeutic option for SS patients' symptoms relief.

DETAILED DESCRIPTION:
The present study is designed as a 24-month, single centre, double-blind, randomized, controlled, two-arm clinical trial (acupuncture and control). The research will be conducted following the CONSORT recommendations and the STRICTA extension. The study care protocol will consist in acupuncture or control intervention at the selected acupoints (R6, E6,E2, Ig4, VC24, TA23, B2) for 8 weeks, 20 minutes sessions with 12 weeks of follow up. Complementary clinical approaches (sialometry, sialochemistry, Schirmer test, staining with topical lissamine green), and the questionnaires (OHIP-14, Eular Sjögren's Syndrome Patient Reported Index (ESSPRI), Xerostomia Inventory, ocular surface disease index (OSDI) will be performed in weeks 1, 8 and 12. The control group will consist of superficial acupuncture, or placebo, or sham. After all interventions and evaluation methods completed, data will be analyzed for their distribution and homogeneity in order to choose the most appropriate statistical test.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old, both genres, who consent to participate of the study
* Patients who were diagnosed with SJ according to the criteria of the American College of Rheumatology and the European League against Rheumatism

Exclusion Criteria:

* Patients who have undergone head and neck radiation therapy;
* Patients with a history of neoplasias and salivary gland infections;
* Patients with acquired immunodeficiency virus infection, sarcoidosis, viral hepatitis, diabetes mellitus and smokers;
* Patients with inability to undergo total saliva collection by established techniques;
* Patients who can not attend regular acupuncture sessions;
* Patients who had a change in the dosage of medications in use within 6 weeks before the start of the study.
* Patients who received acupuncture therapy up to 6 weeks prior to the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Changes from baseline Oral Health Impact Profile (OHIP-14) score at 2 and 3 months. | Before (baseline), immediately after and 1 month after acupuncture treatment.
  Instrument of data collection which comprises of 14 questions with two questions each under seven domains. The domains include; functional limitation,physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. Responses to the questions are based on a Likert scale which ranged from 0- "never" to 4- "always".
Changes from baseline Xerostomia Inventory score at at 2 and 3 months. | Before (baseline), immediately after and 1 month after acupuncture treatment.
  It is an 11-item questionnaire that covers both experiential and behavioral aspects of xerostomia. Scores to the 11 items are summated, providing a single score representing the subjective severity of xerostomia.
Changes from baseline The Challacombe scale at at 2 and 3 months. | Before (baseline), immediately after and 1 month after acupuncture treatment.
  The purpose of this scale is to be able to visually identify and quantify whether your patient has xerostomia (dry mouth)
Changes from baseline EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) at 2 and 3 months. | Before (baseline), immediately after and 1 month after acupuncture treatment.
  There is a 0-10 numerical scale for each of the four domains, dryness, discomfort (including pain), global fatigue and mental fatigue
Changes from baseline Ocular Surface Disease Index (OSDI) at 2 and 3 months. | Before (baseline), immediately after and 1 month after acupuncture treatment.
  This 12-item questionnaire assesses dry eye symptoms and the effects it has on vision-related function in the past week of the patient's life. The questionnaire has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on a 0 to 4 scale with 0 corresponding to "none of the time" and 4 corresponding to "all of the time."

SECONDARY OUTCOMES:
Changes from baseline whole unstimulated salivary flow rate at 2 and 3 months. | Before (baseline), immediately after and 1 month after acupuncture treatment.
  Samples of total saliva (saliva resulting from all salivary glands) will be collected between 8:00 am and 11:00 am, and evaluation of salivary flow will be determined by means of expectoration of saliva in graduated tube of 15 mL for a period of 15 minutes, and the volume obtained will be calculated.
Changes from baseline Schirmer test scores at 2 and 3 months. | Before (baseline), immediately after and 1 month after acupuncture treatment.
  Objective reflection to the lacrimal gland. Schirmer's test uses paper strips inserted into the eye for several minutes to measure the production of tears
Changes from baseline ocular surface staining at 2 and 3 months. | Before (baseline), immediately after and 1 month after acupuncture treatment.
  This is a test that uses orange dye (fluorescein) and a blue light to detect foreign bodies in the eye. This test can also detect damage to the cornea.

CONTACTS AND LOCATIONS:
Overall Officials: Jaciara M Gomes-Silva, DDS, PhD, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil.; Maria Cristina Borsato, DDS, PhD, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil.; Eduardo Melani Rocha, DDS, PhD, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil.; Fabiola R Oliveira, DDS, PhD, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil.; Maria da Conceição P Saraiva, DDS, PhD, Study Chair — University of São Paulo, Ribeirão Preto, SP, Brazil.
Locations (1):
- School of Dentistry of Ribeirão Preto, University of São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Deng G, Hou BL, Holodny AI, Cassileth BR. Functional magnetic resonance imaging (fMRI) changes and saliva production associated with acupuncture at LI-2 acupuncture point: a randomized controlled study. BMC Complement Altern Med. 2008 Jul 7;8:37. doi: 10.1186/1472-6882-8-37. PMID 18606019
- [Background] Jiang Q, Zhang H, Pang R, Chen J, Liu Z, Zhou X. Acupuncture for Primary Sjogren Syndrome (pSS) on symptomatic improvements: study protocol for a randomized controlled trial. BMC Complement Altern Med. 2017 Jan 19;17(1):61. doi: 10.1186/s12906-017-1559-9. PMID 28103850
- [Background] Hackett KL, Deane KH, Strassheim V, Deary V, Rapley T, Newton JL, Ng WF. A systematic review of non-pharmacological interventions for primary Sjogren's syndrome. Rheumatology (Oxford). 2015 Nov;54(11):2025-32. doi: 10.1093/rheumatology/kev227. Epub 2015 Jun 30. PMID 26135587
- [Background] Assy Z, Brand HS. A systematic review of the effects of acupuncture on xerostomia and hyposalivation. BMC Complement Altern Med. 2018 Feb 13;18(1):57. doi: 10.1186/s12906-018-2124-x. PMID 29439690
- [Background] Hu WL, Wu PC, Pan LY, Yu HJ, Pan CC, Hung YC. Effect of laser acupuncture on dry eye: A study protocol for a 2-center randomized controlled trial. Medicine (Baltimore). 2018 Jun;97(22):e10875. doi: 10.1097/MD.0000000000010875. PMID 29851803
- [Background] Kim BH, Kim MH, Kang SH, Nam HJ. Optimizing acupuncture treatment for dry eye syndrome: a systematic review. BMC Complement Altern Med. 2018 May 3;18(1):145. doi: 10.1186/s12906-018-2202-0. PMID 29724255